CLINICAL TRIAL: NCT00823225
Title: Low Dose Urokinase Therapy in Patients With Diabetic Foot Syndrome and Critical Limb Ischemia Versus Conventional Standard Therapy
Brief Title: Urokinase Therapy in Patients With Diabetic Foot Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient recruitment of study patients
Sponsor: medac GmbH (Industry)
Responsible Party: Prof.Dr.med. S. Schellong, Städtisches Krankenhaus Dresden-Friedrichstadt, Friedrichstr. 41, 01067 Dresden, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC-UK.3/AVK; EudraCT number 2007-005916-15
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Diabetic Foot; Arterial Occlusive Disease; Ischemia
Keywords: Diabetes; urokinase; ulcer healing; major amputation; survival
MeSH Terms: conditions — Diabetic Foot; Arterial Occlusive Diseases; Ischemia; Diabetes Mellitus | interventions — Standard of Care; Urokinase-Type Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Standard therapy (Other)
  Interventions: Procedure: standard therapy
- B: Urokinase (Experimental)
  Interventions: Drug: Urokinase

INTERVENTIONS:
Procedure: standard therapy — wound debridement, moist wound dressing
  Arms: A: Standard therapy
Drug: Urokinase — Daily infusion up to 21 applications, dose dependent on fibrinogen level:
  > 2,5g/l 1 000 000 IU, < 2,5g/l 500 000 IU
  Arms: B: Urokinase

SUMMARY:
The purpose of this study is to determine whether the additional therapy with low dose urokinase is more effective than only a conventional standard therapy concerning ulcer-healing, rate of major amputation and survival.

DETAILED DESCRIPTION:
Patients with diabetic foot ulceration and critical limb ischemia have a high risk of major amputation, especially if limbs can not be revascularized. Urokinase is effective in critical limb ischemia by lowering fibrinogen and might improve outcomes. The effect and safety of urokinase treatment was investigated in a phase II clinical trial. Based on the results this trial was planned to investigate the effect and safety of an additional therapy with urokinase versus a single conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with angiopathic or angioneuropathic diabetic foot syndrome and criticial limb ischemia
* No surgical or interventional treatment option
* No healing tendency of ulcerations despite of antibiosis and wound debridement after two-week treatment
* Fibrinogen > 4.0 g/l
* No previous major amputation

Exclusion Criteria:

* Prior treatment of the current ulceration with urokinase
* Need for dialysis and/or creatinine-clearance < 20ml/min
* INR > 1,5 at screening
* Any kind of cerebral event within 3 months prior inclusion
* Proliferative retinopathy
* Uncontrolled hypertension
* Hemorraghic diathesis
* Gastrointestinal bleeding
* Pregnancy
* No compliance and/or participation in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Major amputation free survival | Within twelve months after randomisation

SECONDARY OUTCOMES:
Total survival, major amputation rate, rate of complete ulcer healing, rate of adverse events | Within twelve month after randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Schellong, MD, Principal Investigator — Krankenhaus Dresden-Friedrichstadt, Germany
Locations (6):
- Germany (6):
  - Franziskus Krankenhaus, Berlin
  - Klinikum Dortmund Nord GmbH, Dortmund
  - Krankenhaus Dresden-Neustadt, Dresden
  - Universitätsklinik, Dresden
  - Weißeritztal-Kliniken GmbH, Freital
  - Klinikum Karlsbad Langensteinbach, Karlsbad